CLINICAL TRIAL: NCT06460428
Title: The Effect of Online Interactive Education Provided to Couples Applying for Wedding Via Web-Based Platform on Fertility Awareness
Brief Title: Online Interactive Video Developed for Fertility Awareness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GaziU-Hem-ŞYS-08
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Fertility Awareness
Keywords: Fertility awareness, Pre-wedding period, Web-based education

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental study with a pretest-posttest control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to prevent selection bias and to ensure similarity between groups; simple randomization will be used to assign the couples in the sample group to the experimental and control groups.
  In this study, researcher and participant blinding will not be performed. Because the researcher will do the intervention himself/herself and placebo will not be used in the intervention.
  Data collection forms to prevent detection bias will be applied online through Google Forms® independently of the researcher.
  The data obtained from the research to prevent reporting bias will be transferred to the SPSS program by an independent researcher. Analysis of the data will also be done by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: 1. group (Experimental): Couples in the pre-wedding period will receive information about fertility awareness with the developed interactive video
  Interventions: Behavioral: Interactive video usage
- No Intervention: 2. Group (No Intervention): Control Group (non- education): No intervention will be made

INTERVENTIONS:
Behavioral: Interactive video usage — The implementation of the research was carried out in two stages. In the first stage, interactive videos were created, in the second stage, the experimental group was trained with interactive videos, and no intervention was made to the control group.
  Arms: Active Comparator: 1. group

SUMMARY:
The main purpose of this research is to evaluate the effect of online interactive education provided to newly married couples via a web-based platform on fertility awareness.Since fertility awareness is a relatively new field of research, there are limited studies on this subject. These studies are generally given to women. But the concept of fertility in question concerns not only women but also men.The study conducted via web-based online interactive video developed to raise awareness about fertility; It is thought that raising the awareness of newly married couples, regulating fertility, and including men in this issue are important for public health and will set an example for future studies.The positive outcomes from Webb-based online videos will enable the application to be used on national and international platforms.

DETAILED DESCRIPTION:
Fertility awareness is an understanding that enables individuals to be informed about their reproductive health, fertility cycle and reproductive systems. This understanding enables individuals to gain awareness about their reproductive capacity, fertile periods, sexual health and family planning. Increasing fertility awareness will contribute to increasing the general health and welfare of both individuals and society.Since fertility awareness is a relatively new field of research, there are limited studies on this subject. These studies are generally aimed at women. However, the concept of fertility in question concerns not only women but also men. Individuals who are about to get married have a very important place in processing fertility awareness. The high interest in premarital sexuality, labor and birth, and the motivation for education on this subject make it important for it to be considered as a "missed opportunity" during the application period for marriage procedures. No study has been found in the literature on the development of fertility awareness, including the period of application for marriage. It is expected that the research to be conducted will contribute to the literature in terms of filling the gap in this field, obtaining new data and guiding new strategies to be created.Since information about fertility mostly involves confidential issues, individuals cannot talk about this subject comfortably and cannot obtain information. At the same time, the formation and development of fertility awareness includes individual behavioral changes. Therefore, the education given to couples can be used continuously and in the long term. For such reasons, people prefer online educational materials. Online training helps people feel more comfortable, remain anonymous while learning about these topics, and progress according to their learning pace. Web-based platforms contribute to individuals' awareness of fertility awareness and making healthy decisions by being an effective tool in reaching large audiences, being low-cost and easily accessible, and offering independence of time and place.

The research is a pretest-posttest randomized controlled experimental study conducted to evaluate the effect of online interactive education given to couples applying for marriage via a web-based platform on fertility awareness. It is planned to be conducted with 70 couples (experimental group: 35 couples, control group: 35 couples) who applied to the marriage office of Kecioren Municipality. Couples who apply to the registry office and agree to participate in the research will be asked to fill out the Introductory Information Form, Fertility Awareness Scale and Fertility Health Information Scale. Afterwards, these couples will be randomized and assigned to experimental and control groups. Training content will be created for the couples assigned to the experimental group.After receiving expert opinions on the training content, interactive videos will be prepared via the website httpp://h5ptr.org/. In these interactive videos; It is planned to have 4 modules: anatomy and physiology of the male and female reproductive system, family planning method based on fertility awareness, modern family planning method and factors affecting fertility. While watching these videos, there will be fill-in-the-blank, true-false, and multiple choice questions at certain parts of the videos. If participants answer the questions incorrectly, they will be directed to the section in the video where the answer to the question is found. A website will be prepared for couples to access these interactive videos. The address of this website and the educational content will be sent as an online file to the couples' phones or e-mails. Participants will be asked to complete these trainings within 2 weeks at most and before the wedding. After the training is completed and 1 month after the wedding, participants will fill out the Fertility Awareness Scale and Fertility Health Information Scale via an online survey (Google Forms®). No intervention will be made to the participants in the control group. Before the wedding and one month after the wedding, participants will fill out the Fertility Awareness Scale and Fertility Health Information Scale via an online survey (Google Forms®). In this way, the effect of the online interactive training we have implemented on the fertility awareness of couples applying for marriage will be evaluated. After the data collection tools are completed, the analysis and reporting part will be carried out. Statistical analyzes will be performed using Statistical Package of SocialSciences 27.0 package program. Shapiro-Wilk test, Chi-square test, dependent and independent group t test, Mann Whitney U test will be used in the analysis.

In the research conducted through web-based online interactive video developed to raise awareness about fertility; It is thought that raising the awareness of newly married couples, regulating fertility and including men in this issue are important for public health and will set an example for future studies. The positive results obtained from web-based online videos will enable the application to be used on national and international platforms.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having applied for official marriage
* First marriage
* Must be at least a primary school graduate

Exclusion Criteria:

* Not knowing Turkish
* Having any communication problems (mental, auditory, visual, etc.)
* Having previously received preconception training/care
* There is less than 2 weeks between the marriage ceremony and the marriage application date.

For female participants;

* Having had previous pregnancy or birth experience
* Having been diagnosed with menopause

Criteria for Exclusion from the Sample During the Study:

* Inaccessibility of the study at any stage
* Wanting to leave work
* Completion of training
* Not completing post-tests

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-24 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fertility Awareness Scale | 3 months
  Fertility Awareness Scale is a 19-item, five-point Likert type (1-Never, 2-Rarely, 3-Sometimes, 4-Often, 5-Always), two-dimensional scale: Body Awareness Sub-Dimension 7,9,10, 11,12,13,15,17,18,19 (10 items) and Cognitive Awareness Sub-Dimension 1,2,3,4,5,6,8,14,16 (9 items). There are no reverse items in the scale. The lowest score that can be obtained in the total of the Fertility Awareness Scale is 19 and the highest score is 95. As the total score from the Fertility Awareness Scale increases, the level of awareness increases. If the total score is between 19-43, awareness is classified as low, between 44-69, awareness is classified as medium, and between 70-95, awareness is classified as high level.
Fertility Health Information Scale | 3 months
  Fertility Health Information Scale includes biological information regarding gender-specific reproductive health (menstrual cycle, sperm survival and quality, ability to have an erection), non-modifiable (age) and modifiable (lifestyle choices such as weight, stress, marijuana and cigarette use). /exposure) related to healthy fertility, It includes statements about factors such as stress, caffeine, diet, exercise, sleep habits, etc.). The scale consists of 30 items and has a single-factor structure. Responses to the items related to the scale are on a five-point Likert type (5-definitely yes; 4-probably yes; 3-undecided; 2-probably no; 1-definitely no). Those who choose "definitely yes" or "probably yes" are considered correct. In the evaluation, item 20 is reverse coded. Scores between 0 and 30 points can be obtained from the scale, and as the score increases, knowledge increases.

CONTACTS AND LOCATIONS:
Overall Officials: Şengül Yaman Sözbir, Study Director — Head of Department of Obstetrics and Gynecology Nursing, Gazi University

IPD SHARING:
Plan to Share IPD: No